CLINICAL TRIAL: NCT01293214
Title: Vascularized Composite Allotransplantation for Multiple Extremity Amputations
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Simon George Talbot, Director, Upper Extremity Transplant Program, Brigham and Women's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2012P000073
Record Dates: First submitted 2011-02-09; First posted 2011-02-10 (Estimated); Last update posted 2025-02-05 (Actual); Status verified 2024-08

CONDITIONS: Limb Amputation; Extremity Amputation
Keywords: limb transplantation; limb allotransplantation; hand transplantation; hand allotransplantation; hand amputation; leg transplantation
MeSH Terms: interventions — Vascularized Composite Allotransplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | US Export: No

ARMS (1):
- Transplantation (Experimental): Subjects will undergo single or multiple limb transplantation
  Interventions: Procedure: Limb transplantation

INTERVENTIONS:
Procedure: Limb transplantation
  Other Names: vascularized composite allotransplantation

SUMMARY:
Limb transplantation surgery is the transfer of one or more limbs from a deceased human donor to a patient with single or multiple limb amputation. Hand transplantation is an innovative reconstructive procedure that has the potential to significantly improve the lives of hand amputees. The purpose of this study is to develop the best practices for multiple limb transplantation that will improve the outcomes of future limb transplant recipients.

DETAILED DESCRIPTION:
Limb transplantation surgery, the transfer of the limb(s) from a deceased human donor to a patient with amputation of one or more limbss, is an experimental reconstructive procedure that has the potential to significantly improve the lives of amputees.

Limb transplantation is similar to face transplantation in that the tissues transplanted include skin, tendons, muscles, ligaments, bones and blood vessels. The transplant team at Brigham and Women's Hospital includes a wide variety of medical and surgical specialties. The team hopes to build upon the success of their first face transplantation to provide amputee patients with the significant benefits of limb transplantation.

Toward this goal, BWH is actively seeking qualified candidates for the limb transplant research study. We will be studying a small group of people to learn more about:

* How to advance the science of limb transplantation
* How to support and limit transplant rejection issues
* How people do after limb transplantation

We describe limb transplant surgery as a life-giving procedure because it has the potential to dramatically improve, that is to restore, both a patient's mental and physical health and his/her ability to function and integrate in society. However, as with any other type of organ transplantation, this improvement will require the patient to make a lifetime commitment to taking medications that suppress the body's immune system.

Conventional reconstruction methods are always considered first, but they may provide less than optimal results for certain patients. There are many sophisticated prostheses that satisfactorily replace the basic function of a missing limb. However, replacing limbs (in whole or in part) with prosthetics remains suboptimal in that prostheses do not provide sensation and do not have a natural appearance. Limbtransplant surgery, however, has the potential to deliver these desired functional and aesthetic benefits. Functionally, limb transplant surgery can provide a patient with new limbs that, after extensive rehabilitation, allow him/her to perform daily activities and, in most cases, return to work. Furthermore, the ability to restore a near-normal aesthetic appearance of the limb(s) can lead to tremendous psychological benefits, including elevated confidence and mood.

From the time we begin our search for a qualified limb transplant recipient to the continuing care we provide following surgery, a significant amount of time, expertise and attentiveness is contributed toward making the procedure a progressive success. Limb transplant candidates go through an extensive screening process that is likely to last several months. This screening includes a psychiatric and social support evaluation and a series of imaging tests to help determine a patient's physical and mental readiness for the procedure. If, upon completion of the screening process, it is determined that a patient is a suitable candidate, we will place the patient on a transplant waiting list. We will then begin working with the New England Organ Bank (NEOB) team to find a donor who matches the recipient's tissue requirements - for example similar age and correct blood type. This search could take many months, and, if a suitable donor is not found within one year, we will speak with the patient to determine whether he/she is willing to continue waiting.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 60 years.
* Single dominant hand or multiple limb amputation.
* Time elapsed since amputation more than 6 months but less than 15 years.
* Patient has tried prosthesis without success.
* Level of amputation anywhere from the wrist (or ankle) joint to just below the shoulder (or hip) joint, which should be functional.
* Signed written informed consent.
* Willing to complete psychological and social evaluations.
* Willing to take immunosuppressants - drugs that help prevent rejection of the transplant - for life.
* Willing to comply with extensive post-transplant rehabilitation for a minimum of two years.
* Willing to return for follow-up visits as determined by the treating physician.
* Willing to receive standard vaccinations prior to the transplant, such as influenza and hepatitis B.

Exclusion Criteria:

* Single, non-dominant hand amputees.
* Active malignancy.
* High risk of return of malignancy.
* History of persistent non-compliance.
* Findings of psychological evaluation that indicate inability to comply with physician's orders or mental instability.
* Any diagnosis that puts the subject at risk from limb transplant surgery or life-long immune suppression.
* Inability to ensure adequate follow-up of post-transplant care and immune suppression.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Estimated)
Dates: Start 2010-02-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Outcomes of limb transplantation | Subjects will be followed for 18 months after transplantation
  We will undertake an objective evaluation of the results of limb transplantation in an "outcome-oriented" study

SECONDARY OUTCOMES:
Efficacy and optimization of the immune suppression protocol | 18 months
  We will evaluate the risks of rejection or likelihood of tolerance induction by measuring specific parameters in the blood or tissue, including: Serum alloantibodies concentration, numbers/phenotype of specific T cell alloreactivity in the peripheral blood, phenotypic characterization of graft infiltrating cells and local gene expression of cells and cytokines.

CONTACTS AND LOCATIONS:
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Background] Pomahac B, Aflaki P. Composite tissue transplantation: a new era in transplantation surgery. Eplasty. 2010 Sep 15;10:e58. PMID 20862294
- [Background] Bueno E, Benjamin MJ, Sisk G, Sampson CE, Carty M, Pribaz JJ, Pomahac B, Talbot SG. Rehabilitation following hand transplantation. Hand (N Y). 2014 Mar;9(1):9-15. doi: 10.1007/s11552-013-9568-8. PMID 24570631
- [Background] George E, Mitsouras D, Kumamaru KK, Shah N, Smith SE, Schultz K, Deaver PM, Mullen KM, Steigner ML, Gravereaux EC, Demehri S, Bueno EM, Talbot SG, Pomahac B, Rybicki FJ. Upper extremity composite tissue allotransplantation imaging. Eplasty. 2013 Jul 16;13:e38. eCollection 2013. PMID 23943677
- [Background] Carty MJ, Zuker R, Cavadas P, Pribaz JJ, Talbot SG, Pomahac B. The case for lower extremity allotransplantation. Plast Reconstr Surg. 2013 Jun;131(6):1272-1277. doi: 10.1097/PRS.0b013e31828bd1a5. PMID 23416434
- [Derived] Borges TJ, Abarzua P, Gassen RB, Kollar B, Lima-Filho M, Aoyama BT, Gluhova D, Clark RA, Islam SA, Pomahac B, Murphy GF, Lian CG, Talbot SG, Riella LV. T cell-attracting CCL18 chemokine is a dominant rejection signal during limb transplantation. Cell Rep Med. 2022 Mar 15;3(3):100559. doi: 10.1016/j.xcrm.2022.100559. eCollection 2022 Mar 15. PMID 35492875
- See also: Study's official webpage — https://www.brighamandwomens.org/surgery/plastic-surgery/restorative-surgery/hand-arm-transplant-surgery